CLINICAL TRIAL: NCT01896388
Title: Ifenprodil Tartrate Treatment of Adolescents With Post-traumatic Stress Disorder: a Double-blind, Placebo-controlled Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chiba University (Other)
Responsible Party: Principal Investigator, Tsuyoshi Sasaki, Tsuyoshi Sasaki, Clinical Associate Professor, Chiba University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G25013
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Posttraumatic Stress Disorders
Keywords: PTSD/ifenprodil
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — ifenprodil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ifenprodil Tartrate (Active Comparator): Oral Administration of Ifenprodil Tartrate 40mg/day (20mg After breakfast, 20mg After supper)
  Interventions: Drug: Ifenprodil Tartrate
- Placebo (Placebo Comparator): Oral Administration of Placebo (After breakfast, After supper)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ifenprodil Tartrate
  Arms: Ifenprodil Tartrate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Accumulating evidence suggests a key role of the N-methyl-D-aspartate (NMDA) receptor in the pathophysiology of post-traumatic stress disorder (PTSD). Recent studies suggest that the NMDA receptor antagonist ifenprodil tartrate may be a potential therapeutic drug for PTSD. The purpose of this study is to confirm whether ifenprodil tartrate is effective in the treatment of adolescents PTSD patients. If ifenprodil tartrate is effective in these patients, this study contributes to the development of novel therapeutic drugs for PTSD.

ELIGIBILITY:
[Inclusion Criteria]

1. Diagnosis of PTSD based on DSM-IV-TR criteria.
2. Score of 25 or higher on the IES-R.
3. currently is an outpatient at Chiba University Hospital Department of Psychiatry or Child Psychiatry .
4. currently receiving no medications for PTSD treatment with any of the following medications : Antidepressants (SSRI ; Fluvoxamine, Paroxetine, Sertraline, Escitalopram, SNRI ; Milnacipran, Duloxetine, NaSSa; Mirtazapine), Mood stabilizers (Lithium, Sodium Valproate, Carbamazepine, Lamotrigine), Atypical antipsychotics (Risperidone, Olanzapine, Quetiapine, Perospirone, Aripiprazole, Blonanserin, Paliperidone) .
5. Ages 13 - 18, male or female
6. be stable on any medications for PTSD treatment they may be taking for the previous 4 weeks prior to enrollment in this study.
7. Provision of written informed consent by patients and parents or guardian.
8. must be able to swallow powdered medicine.

[Exclusion Criteria]

1. History of allergic reaction or hypersensitivity to Ifenprodil Tartrate.
2. Patients who have not stopped bleeding after intracranial hemorrhage.
3. Patients who have not been informed of having the disease at the time of informed consent.
4. Diagnosis of any of the following diseases based on the DSM-IV-TR criteria. Mental Retardation, Pervasive Developmental Disorders, Attention-Deficit / Hyperactivity Disorder, Schizophrenia and Other Psychotic Disorders, Delirium, Dementia, and Amnestic and Other Cognitive Disorders, Substance-Related Disorders (except Caffeine-Related Disorders, Nicotine-Related Disorders) .
5. Somatic disorder which requires severe body management or severe meal management.
6. receiving treatment, with antidepressants, mood stabilizers, and atypical antipsychotics other than those of the inclusion criteria #4, within 4 weeks prior to enrollment in this study.
7. receiving treatment with the following N-methyl-D-aspartate (NMDA) receptor antagonists: Ketamine hydrochloride, Amantadine hydrochloride, Memantine hydrochloride, dextromethorphan, Methadone) within 4 weeks prior to enrollment in this study.
8. pregnant or nursing, or intending to become pregnant or to start breastfeeding during the study.
9. participating in another clinical trial within 3 months prior to enrollment into this study. (except for observation study without intervention).
10. planning change of treatment because of unstable neurological manifestations or somatic symptoms.
11. History of suicidal ideation within the past year.
12. Other clinically significant reasons for exclusion by investigators.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01-21 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
The Impact of Event Scale-Revised Japanese Version : IES-R-J | Changes from baseline in IES-R-J at 4-weeks
  Evidence includes retest reliability and internal consistency of the IES-R-J. Posttraumatic stress disorder (PTSD) and partial PTSD cases indicated significantly higher scores than non-PTSD cases. The IES-R-J can be a useful self-rating diagnostic instrument particularly for survivors with PTSD symptoms as a clinical concern (PTSD + partial PTSD) by using a 24/25 cutoff in total score. The IES-R-J can be used as a validated instrument in future international comparative research.

SECONDARY OUTCOMES:
Trauma Symptom Checklist for Children Japanese Version : TSCC-J | Changes from baseline in TSCC-J at 4-weeks
  The TSCC allows you to measure posttraumatic stress and related psychological symptomatology in children ages 8-16 years who have experienced traumatic events, such as physical or sexual abuse, major loss, or natural disasters, or who have been a witness to violence.
  The 54-item TSCC includes two validity scales (Underresponse and Hyperresponse), six clinical scales (Anxiety, Depression, Anger, Posttraumatic Stress, Dissociation, and Sexual Concerns), and eight critical items. Profile Forms allow for conversion of raw scores to age- and sex-appropriate T scores and enable you to graph the results.
  The TSCC-A, an alternate 44-item version of the measure, makes no reference to sexual issues.

OTHER OUTCOMES:
Children's Depression Rating Scale-Revised : CDRS-R | Changes from baseline in CDRS-R at 4-weeks
  The CDRS-R is a brief rating scale based on a semi-structured interview with the child (or an adult informant who knows the child well). Designed for 6- to 12-year-olds, and successfully used with adolescents, it can be administered in just 15 to 20 minutes and easily scored in a few minutes more. The interviewer rates 17 symptom areas (including those that serve as DSM-IV criteria for a diagnosis of depression)
Depression Self-Rating Scale for Children Japanese Version: DSRS-C-J | Changes from baseline in DSRS-C-J at 4-weeks
  DSRS-C-J is easy to use and has a predictive value comparable with that of a psychiatric global rating of depressed appearance and history of depression obtained at interview. There was confirmation that the DSRS-C-J can tap an internal dimension of depression and that children are able to evaluate their feeling states.
Clinical Global Impressions-Post Traumatic Stress Disorder-Improvement : CGI-PTSD-I | Changes from baseline in CGI-PTSD-I at 4-weeks
  The Clinical Global Impression rating scales are commonly used measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders (Guy, W., 1976).
  The Clinical Global Impression - PTSD - Improvement scale (CGI-PTSD-I) is a 7 point scale that requires the clinician to assess how much the PTSD has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Clinical Global Impressions-Post Traumatic Stress Disorder-Severity : CGI-PTSD-S | Changes from baseline in CGI-PTSD-S at 4-weeks
  The Clinical Global Impression rating scales are commonly used measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders (Guy, W., 1976).
  The Clinical Global Impression -PTSD - Severity scale (CGI-PTSD-S) is a 7-point scale that requires the clinician to rate the severity of the PTSD at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.

CONTACTS AND LOCATIONS:
Overall Officials: Masaomi Iyo, MD,PhD, Study Chair — Chairman, Department of Psychiatry, Chiba University Graduate School of Medicine; Nobuhisa Kanahara, MD,PhD, Study Director — Division of Medical Treatment and Rehabilitation, Chiba University Center for Forensic Mental Health; Tasuku Hashimoto, MD.PhD, Study Director — Department of Psychiatry, Chiba University Graduate School of Medicine; Akihiro Shiina, MD,PhD, Study Director — Department of Child Psychiatry, Chiba University Hospital; Tomihisa Niitsu, MD,PhD, Study Director — Research Center for Child Mental Development, Chiba University Graduate School of Medicine
Locations (1):
- Department of Psychiatry, Chiba University School of Medicine Chiba, Chuo-ku, Japan 260-8670, Chiba, Chuo-ku, Japan